CLINICAL TRIAL: NCT05658887
Title: A Double-Blind Randomized Placebo-Controlled Clinical Trial of Preoperative Gabapentin Prior to Vaginal Apical Suspension Prolapse Procedures
Brief Title: Preoperative Gabapentin vs Placebo for Vaginal Prolapse Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Kowalski (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Joseph Kowalski, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202207210
Record Dates: First submitted 2022-12-09; First posted 2022-12-21 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse; Perioperative/Postoperative Complications
Keywords: perioperative pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Postoperative Complications | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Preoperative tylenol, preoperative celecoxib, preoperative gabapentin placebo
  Interventions: Drug: Gabapentin Placebo
- Intervention (Experimental): Preoperative tylenol, preoperative celecoxib, preoperative gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — One dose of preoperative gabapentin 300 mg prior to vaginal apical support procedure
  Other Names: FusePaq Fanatrex; Gabarone; Gralise; Neurontin
  Arms: Intervention
Drug: Gabapentin Placebo — Gabapentin Placebo
  Other Names: FusePaq Fanatrex Placebo; Gabarone Placebo; Gralise Placebo; Neurontin Placebo
  Arms: Placebo

SUMMARY:
This study will recruit women scheduled to undergo vaginal apical suspension surgery (either uterosacral ligament suspension or sacrospinous ligament fixation) with or without other prolapse or anti-incontinence procedures. Participants will be randomized 1:1 to preoperative gabapentin or preoperative placebo (both patients and investigators will be blinded). Note the control group will receive preoperative acetaminophen/celecoxib/placebo and the treatment group will receive preoperative acetaminophen/celecoxib/gabapentin (preoperative acetaminophen/celecoxib are part of our current ERAS protocol). The primary outcome will be postoperative opioid use in the first 24 hours postoperatively measured in morphine milligram equivalents.

DETAILED DESCRIPTION:
Enhanced Recovery after Surgery (ERAS) is an approach to perioperative care that focuses on evidence-based care protocols that emphasize minimizing stress and improving the body's response to stress. These protocols have resulted in a significant decrease in length of stay, complications, and cost in many different surgical specialities. Many of these protocols (including our current gynecology ERAS protocol) include preoperative gabapentin as an intervention to help reduce postoperative pain and postoperative opioid use. Gabapentin is an anticonvulsant medication that is commonly used for chronic neuropathic pain and other chronic pain disorders. The data regarding perioperative use of gabapentin is currently mixed, and the data in gynecology (and especially urogynecology) is limited. Notably gabapentin has been shown to be associated with sedation, respiratory depression, dizziness, and visual disturbances. In 2019, the U.S. Food and Drug Administration issued a warning that serious breathing difficulties may occur in patients using gabapentin with respiratory risk factors.

Pelvic organ prolapse is a common benign condition, and surgery for pelvic organ prolapse is very common. Vaginal apical suspension is one of the most common surgeries for pelvic organ prolapse. There is very limited data on the utility of preoperative gabapentin for vaginal apical suspension surgery.

This study will recruit women scheduled to undergo vaginal apical suspension surgery (either uterosacral ligament suspension or sacrospinous ligament fixation) with or without other prolapse or anti-incontinence procedures. Participants will be randomized 1:1 to preoperative gabapentin or preoperative placebo (both patients and investigators will be blinded). Note the control group will receive preoperative acetaminophen/celecoxib/placebo and the treatment group will receive preoperative acetaminophen/celecoxib/gabapentin (preoperative acetaminophen/celecoxib are part of our current ERAS protocol). The primary outcome will be postoperative opioid use in the first 24 hours postoperatively measured in morphine milligram equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a vaginal apical support procedure (sacrospinous ligament fixation or vaginal uterosacral ligament suspension)
* Female
* Age 18 or higher

Exclusion Criteria:

* Non-English speaking
* Incarcerated
* Cognitive impairment precluding informed consent
* Chronic opioid user
* Chronic gabapentinoid user
* Contraindication to acetaminophen, celecoxib, or gabapentinoids
* Concurrent laparoscopic or abdominal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kowalski, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Smith TW Jr, Wang X, Singer MA, Godellas CV, Vaince FT. Enhanced recovery after surgery: A clinical review of implementation across multiple surgical subspecialties. Am J Surg. 2020 Mar;219(3):530-534. doi: 10.1016/j.amjsurg.2019.11.009. Epub 2019 Nov 16. PMID 31761300
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Altman AD, Robert M, Armbrust R, Fawcett WJ, Nihira M, Jones CN, Tamussino K, Sehouli J, Dowdy SC, Nelson G. Guidelines for vulvar and vaginal surgery: Enhanced Recovery After Surgery Society recommendations. Am J Obstet Gynecol. 2020 Oct;223(4):475-485. doi: 10.1016/j.ajog.2020.07.039. Epub 2020 Jul 24. PMID 32717257
- [Background] Scheib SA, Thomassee M, Kenner JL. Enhanced Recovery after Surgery in Gynecology: A Review of the Literature. J Minim Invasive Gynecol. 2019 Feb;26(2):327-343. doi: 10.1016/j.jmig.2018.12.010. Epub 2018 Dec 20. PMID 30580100
- [Background] Mehr AA, Elmer-Lyon C, Maetzold E, Bradley CS, Kowalski JT. Effect of Enhanced Recovery Protocol on Opioid Use in Pelvic Organ Prolapse Surgery. Female Pelvic Med Reconstr Surg. 2021 Dec 1;27(12):e705-e709. doi: 10.1097/SPV.0000000000001114. PMID 34807884
- [Background] Mathieson S, Lin CC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020 Apr 28;369:m1315. doi: 10.1136/bmj.m1315. No abstract available. PMID 32345589
- [Background] Doleman B, Heinink TP, Read DJ, Faleiro RJ, Lund JN, Williams JP. A systematic review and meta-regression analysis of prophylactic gabapentin for postoperative pain. Anaesthesia. 2015 Oct;70(10):1186-204. doi: 10.1111/anae.13179. Epub 2015 Aug 24. PMID 26300519
- [Background] Rorarius MG, Mennander S, Suominen P, Rintala S, Puura A, Pirhonen R, Salmelin R, Haanpaa M, Kujansuu E, Yli-Hankala A. Gabapentin for the prevention of postoperative pain after vaginal hysterectomy. Pain. 2004 Jul;110(1-2):175-81. doi: 10.1016/j.pain.2004.03.023. PMID 15275765
- [Background] Hah J, Mackey SC, Schmidt P, McCue R, Humphreys K, Trafton J, Efron B, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Carroll I. Effect of Perioperative Gabapentin on Postoperative Pain Resolution and Opioid Cessation in a Mixed Surgical Cohort: A Randomized Clinical Trial. JAMA Surg. 2018 Apr 1;153(4):303-311. doi: 10.1001/jamasurg.2017.4915. PMID 29238824
- [Background] Verret M, Lauzier F, Zarychanski R, Perron C, Savard X, Pinard AM, Leblanc G, Cossi MJ, Neveu X, Turgeon AF; Canadian Perioperative Anesthesia Clinical Trials (PACT) Group. Perioperative Use of Gabapentinoids for the Management of Postoperative Acute Pain: A Systematic Review and Meta-analysis. Anesthesiology. 2020 Aug;133(2):265-279. doi: 10.1097/ALN.0000000000003428. PMID 32667154
- [Background] Huynh TQ, Patel NR, Goldstein ND, Makai GE. Preoperative Gabapentin for Minimally Invasive Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Feb;28(2):237-244.e2. doi: 10.1016/j.jmig.2020.04.040. Epub 2020 May 8. PMID 32389735
- [Background] Weingarten TN, Jacob AK, Njathi CW, Wilson GA, Sprung J. Multimodal Analgesic Protocol and Postanesthesia Respiratory Depression During Phase I Recovery After Total Joint Arthroplasty. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):330-6. doi: 10.1097/AAP.0000000000000257. PMID 25967650
- [Background] Pelvic Organ Prolapse: ACOG Practice Bulletin, Number 214. Obstet Gynecol. 2019 Nov;134(5):e126-e142. doi: 10.1097/AOG.0000000000003519. PMID 31651832
- [Background] Sammarco AG, Swenson CW, Kamdar NS, Kobernik EK, DeLancey JOL, Nallamothu B, Morgan DM. Rate of Pelvic Organ Prolapse Surgery Among Privately Insured Women in the United States, 2010-2013. Obstet Gynecol. 2018 Mar;131(3):484-492. doi: 10.1097/AOG.0000000000002485. PMID 29420405
- [Background] Li ALK, Wadsworth K, Siddiqui NT, Alarab M, McDermott CD, Lemos N, Dawood A, Lovatsis D. Does low-dose gapapentin reduce opioid use postoperatively?: A randomized controlled trial in women undergoing reconstructive pelvic surgery. Int Urogynecol J. 2019 Feb;30(2):211-217. doi: 10.1007/s00192-018-3617-3. Epub 2018 Mar 21. PMID 29564507
- [Background] Committee Opinion No. 750: Perioperative Pathways: Enhanced Recovery After Surgery: Correction. Obstet Gynecol. 2019 Nov;134(5):1121. doi: 10.1097/AOG.0000000000003569. No abstract available. PMID 31651825
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Bolliger M, Kroehnert JA, Molineus F, Kandioler D, Schindl M, Riss P. Experiences with the standardized classification of surgical complications (Clavien-Dindo) in general surgery patients. Eur Surg. 2018;50(6):256-261. doi: 10.1007/s10353-018-0551-z. Epub 2018 Jul 24. PMID 30546385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 people completed informed consent. 3 people withdrew or were disqualified prior to being randomized which is why only 107 were randomized.
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 52 | 55
Completed | 50 | 50
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Preoperative tylenol, preoperative celecoxib, preoperative placebo
  Gabapentin Placebo: Gabapentin Placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [52 to 71] | 67 [62 to 74] | 65 [56.75 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 48 | 49 | 97
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.9 [25.9 to 32.6] | 28.3 [26.1 to 32.4] | 28.5 [25.975 to 32.45]
Vaginal Parity [Median (Inter-Quartile Range); unit: Vaginal Deliveries] | 2 [2 to 3] | 3 [2 to 4] | 2.5 [2 to 3]
Current Tobacco Use [Count of Participants; unit: Participants] | 4 | 8 | 12
Diabetes [Count of Participants; unit: Participants] | 4 | 9 | 13
Prior Hysterectomy [Count of Participants; unit: Participants] | 12 | 13 | 25
Prior Pelvic Organ Prolapse (POP) Surgery [Count of Participants; unit: Participants] | 2 | 2 | 4
Prior Stress Urinary Incontinence (SUI) Surgery [Count of Participants; unit: Participants] | 3 | 1 | 4
Pelvic Organ Prolapse Quantification (POP-Q) Stage [Median (Inter-Quartile Range); unit: Stage] — POP-Q Staging System:
  Stage 0: No prolapse
  Stage 1: The most distal portion of the prolapse is more than 1 cm above the level of the hymen
  Stage 2: The most distal portion of the prolapse is 1 cm or less proximal or distal to the hymen
  Stage 3: The most distal portion of the prolapse protrudes more than 1 cm below the hymen but protrudes no farther than 2 cm less than the total vaginal length
  Stage 4: The most distal portion of the prolapse is within 1 cm of the total vaginal length
  Stage | 2 [2 to 3] | 3 [2 to 3] | 2 [2 to 3]
Vaginal Atrophy [Count of Participants; unit: Participants] | 34 | 43 | 77
Baseline Vaginal Estrogen Use [Count of Participants; unit: Participants] | 15 | 13 | 28
Preoperative Pain Score of 0 [Count of Participants; unit: Participants] — This is the numeric rating scale which ranges from 0 to 10. 0 is no pain and 10 is the worst pain possible.
  Participants | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Use
Description: Total postoperative opioid use in the first 24 hours postop measured in MME (starting when the patient leaves the operating room)
Time Frame: 24 hours after surgery. This includes postoperative opioid use in the hospital AND at home (which is why it is different from outcome measure 3).
Measure: Median (Inter-Quartile Range); unit: MMEs
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
MMEs | 25 [13 to 45] | 20 [8 to 35]

2. Secondary Outcome: Mean Postop Pain Score
Description: Mean postoperative pain score (using the validated numerical rating scale, minimum score 0, maximum score 10, higher scores mean worse pain/worse outcome) while admitted in the hospital. Note: this is the mean score while they were postoperatively but median below is correct because we used the median of each individual's MEAN score (this is addressing the comment #10)
Time Frame: From the time surgery finished to a max of 24 hours after. This was measured by postoperative nursing periodically throughout the postoperative period per standard nursing protocol: usually every hour for the first two hours and then every 4 to 8 hours
Measure: Median (Inter-Quartile Range); unit: Pain Score
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Pain Score | 3.5 [2 to 4.8] | 3.25 [2 to 4.5]

3. Secondary Outcome: Postoperative Opioid Use While Admitted in the Hospital
Description: postoperative opioid use while admitted
Time Frame: After surgery, max of 24 hours. Note that this is only postoperative opioid use in the hospital. Outcome measure 1 is total postoperative opioid use (in the hospital and at home)
Measure: Median (Inter-Quartile Range); unit: MMEs
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
MMEs | 20 [5 to 36] | 16 [5 to 25]

4. Secondary Outcome: Time to Discharge
Description: Admitted time
Time Frame: Total admitted time (from admission to the hospital to discharge)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
minutes | 528 [459 to 678] | 542 [477 to 1394]

5. Secondary Outcome: Number of Patients Who Report Postoperative Dizziness
Description: Patient reported postoperative dizziness
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Participants | 13 | 7

6. Secondary Outcome: Number of Patients Who Report Sedation
Description: Patient reported sedation
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Participants | 4 | 2

7. Secondary Outcome: Number of Patients Who Report Visual Changes
Description: Patient reported visual changes
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Participants | 1 | 1

8. Secondary Outcome: Number of Patients Who Report Postoperative Nausea
Description: Patient reported postoperative nausea and vomiting
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Participants | 14 | 10

9. Secondary Outcome: Number of Patients Who Report Postoperative Pain Adequacy
Description: Patient reported postoperative pain adequacy
Time Frame: 24 hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Participants | 40 | 41

10. Secondary Outcome: Morphine Milligram Equivalents (MMEs) of Preoperative and Intraoperative Opioids
Description: Amount of opioids (in MMEs) given before and during the surgery
Time Frame: Preop period to the end of the surgery (any opioids given to the patient from arrival in the hospital to the end of the surgery), on average 5 hours
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents (MMEs)
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Morphine milligram equivalents (MMEs) | 46 [42 to 74] | 40 [34 to 55]

11. Secondary Outcome: Estimated Blood Loss
Time Frame: During the surgery (from surgery start time to surgery end time, this was assessed at the end of the surgery while in the OR), on average 150 minutes
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
mL | 25 [0 to 75] | 50 [10 to 50]

12. Secondary Outcome: Surgery Length
Time Frame: During surgery
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 50 | 50
Minutes | 152 [127 to 170] | 147 [110 to 165]

ADVERSE EVENTS:
Time Frame: 36 hours after surgery
Arm/Group | Placebo | Intervention
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 21/50 | 16/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | Intervention (N=50)
Participant Reported Dizziness (Nervous system disorders) | 13 | 7
Patient Reported Sedation (Nervous system disorders) | 4 | 2
Patient Reported Visual Changes (Nervous system disorders) | 1 | 1
Patient Reported Nausea (Gastrointestinal disorders) | 14 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05658887/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT05658887/ICF_004.pdf